CLINICAL TRIAL: NCT00256997
Title: Pragmatic Randomized Trial of Risperdal Consta Versus Oral Atypical Antipsychotics in Poorly Adherent Subjects With Schizophrenia in a Routine Care Setting
Brief Title: A Study of Risperidone Long-Acting Injection Versus Oral Antipsychotics in Schizophrenia Participants With a History of Being Poorly Compliant With Taking Their Medication
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit number of planned patients
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006016; RISSCH4055
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2013-10-07 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal Consta
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone long-acting injection (LAI) (Experimental): Risperidone LAI 25 milligram (mg), 37.5 mg or 50 mg intramuscular (injection of a substance into a muscle) injection will be administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic will also be administered in the first 3 weeks following the dose increase. Duration of treatment will be 24 months.
  Interventions: Drug: Risperidone long-acting injection (LAI)
- Oral atypical Antipsychotic (Active Comparator): Oral atypical antipsychotic will be administered as per local label practice for 24 months. Participants will be switched to another atypical oral therapy as per Investigator's discretion.
  Interventions: Drug: Oral atypical Antipsychotic

INTERVENTIONS:
Drug: Risperidone long-acting injection (LAI) — Risperidone LAI 25 milligram (mg), 37.5 mg or 50 mg intramuscular (injection of a substance into a muscle) injection will be administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic will also be administered in the first 3 weeks following the dose increase. Duration of treatment will be 24 months.
  Arms: Risperidone long-acting injection (LAI)
Drug: Oral atypical Antipsychotic — Oral atypical antipsychotic will be administered as per local label practice for 24 months. Participants will be switched to another atypical oral therapy as per Investigator's discretion.
  Arms: Oral atypical Antipsychotic

SUMMARY:
The purpose of this study is to evaluate risperidone long-acting injection (an antipsychotic medication) versus oral antipsychotics in schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) participants with a history of being poorly compliant with taking their medication.

DETAILED DESCRIPTION:
This is a Phase 4, an open-label (all people know the identity of the intervention), multi-country and multi-centric (conducted in more than one center) study of risperidone long-acting formulation versus oral (having to do with the mouth) atypical antipsychotics in participants with a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text revision ( DSM-IV TR) diagnosis of schizophrenia currently being treated with oral antipsychotic medication. The duration of this study will be 2 years. All the eligible participants will be randomly assigned to an oral atypical antipsychotic (risperidone, olanzapine, quetiapine, and where commercially available, aripiprazole and amisulpride) or to risperidone long-acting formulation. For risperidone long-acting formulation participants, study medication will be administered by intramuscular (into the muscle) injection every 2 weeks at doses of 25, 37.5 or 50 milligram (mg). Oral supplementation with the current oral atypical antipsychotic is required for the first 3 weeks following the initial injection and dose increase. Dose increase can be made as per product labeling. The primary measure of effectiveness is the reduction in the percentage of participants experiencing a clinical exacerbation after being in the study for 3 months. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) as per Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text revision (DSM-IV TR)- Have had at least 2 hospitalizations or 2 clinical worsening of symptoms, over the past 2 years because of deteriorating adherence - Is currently receiving treatment with an antipsychotic per local product label guidelines, and has a history in the last 5 years of a satisfactory response (minimum of 6 weeks) to oral antipsychotics (excluding clozapine) - On monotherapy antipsychotic treatment as per local product label guidelines, at Baseline -Female participants must be surgically sterile, or practicing an effective method of birth control before entry and throughout the study, and have a negative urine pregnancy test at screening before study entry Exclusion Criteria: - Participants with a primary DSM-IV TR Axis I diagnosis other than schizophrenia - Female participants who are currently pregnant or breastfeeding or planning a pregnancy within 2 years of trial start - Have a serious, unstable and untreated medical illnesses, such as vascular or cardiovascular disease, history of liver or kidney disease, significant cardiac (having to do with the heart), pulmonary (having to do with the lungs), gastrointestinal, endocrine, neurological (pertaining to the nervous system) or metabolic disturbances - At significant risk of suicide or violence at study start - Evidence of substance dependence (except for nicotine and caffeine dependence) according to DSM-IV TR criteria diagnosed in the last month prior to entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (44):
- Australia (5):
  - Dandenong
  - Frankston
  - Mount Claremont
  - Newcastle
  - Southport
- Canada (15):
  - Calgary, Alberta
  - Bathurst, New Brunswick
  - Kentville, Nova Scotia
  - Sydney, Nova Scotia
  - Greater Sudbury, Ontario
  - Kingston, Ontario
  - Mississauga, Ontario
  - Beauport, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Georges, Quebec
  - Battleford, Saskatchewan
  - Prince Albert, Saskatchewan
  - Montreal
  - Saint John
- Ireland (3):
  - Co.Mayo
  - Dublin
  - Mullingar
- United Kingdom (21):
  - Birmingham
  - Boston
  - Bristol
  - Burnley
  - Darwen
  - Devon
  - Grantham
  - Leicester
  - Lincoln
  - London
  - Morpeth
  - Newcastle upon Tyne
  - Northampton
  - Nottingham
  - Preston
  - Stamford
  - Stockton-Upon-Tees
  - Swansea
  - Teignmouth
  - Wallsend
  - Weston-super-Mare

REFERENCES:
- See also: Pragmatic randomized trial of Risperdal Consta versus oral atypical antipsychotics in poorly adherent subjects with schizophrenia in a routine care setting. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=367&filename=CR006016_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Long-Acting Injection (LAI): Risperidone LAI 25 milligram (mg), 37.5 mg or 50 mg intramuscular (injection of a substance into a muscle) injection was administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic was also administered in the first 3 weeks following the dose increase. Duration of treatment was 24 months.
- Oral Atypical Antipsychotic: Oral atypical antipsychotic was administered as per local label practice for 24 months. Participants switched to another atypical oral therapy as per Investigator's discretion.
Period: Overall Study
Arm/Group | Risperidone Long-Acting Injection (LAI) | Oral Atypical Antipsychotic
Started | 81 | 86
Treated | 79 | 86
Completed | 33 | 31
Not Completed | 48 | 55
Not completed — Protocol Violation | 1 | 4
Not completed — Lack of Efficacy | 1 | 4
Not completed — Death | 2 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 13 | 3
Not completed — Started but not treated | 2 | 0
Not completed — Other | 5 | 8
Not completed — End of Study (As Per Sponsor) | 12 | 24
Not completed — Participant Non-compliant | 3 | 6
Not completed — Investigator Withdrew Participant | 2 | 1

BASELINE CHARACTERISTICS:
Population: Out of a total of 167 participants, Baseline data was available for only 165 participants who were included in intent to treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone Long-Acting Injection (LAI) | Oral Atypical Antipsychotic | Total
Number analyzed (Participants) | 79 | 86 | 165
Age Continuous [Mean (Standard Deviation); unit: Years] — Out of a total of 167 participants, Baseline characteristic (Age) was available for only 165 participants who were included in intent to treat (ITT) population.
  Years | 37.4 (12.46) | 38.9 (10.9) | 38.2 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 167 participants, Baseline characteristic (Gender) was available for only 165 participants who were included in intent to treat (ITT) population.
  Participants
    Female | 23 | 23 | 46
    Male | 56 | 63 | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Clinical Exacerbation From Month 3 Post-Randomization
Description: Clinical exacerbation is defined as hospitalization because of participant's schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, delusions, hallucinations, and self withdrawal) or requiring change from current antipsychotic or initiation of adjunctive antipsychotic, 2-point worsening in Clinical Global Impression of Severity (CGI-S) or emergency room visit, deliberate self-injury, emergence of clinically significant suicidal ideation, utilization of treatment team services, violent behavior, requiring an increase in dose of existing antipsychotic as a result of poor symptom control.
Time Frame: Month 3 up to Month 24
Population: Intent-to-treat (ITT) population included all participants who received medication with at least one post-baseline effectiveness measure. This study was stopped due to futility; care must be exercised in any interpretation of utilization of these data.
Measure: Number; unit: Percentage of participants
Arm/Group | Risperidone Long-Acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 86
Percentage of participants | 48.1 | 43.0
Statistical Analysis 1: Comparison: Risperidone Long-Acting Injection (LAI) vs Oral Atypical Antipsychotic; Test type: Superiority or Other; p = 0.5498, Cox proportional hazard model — P-value was calculated by Cox proportional hazard model stratified for positive and negative symptom scale

2. Secondary Outcome: Percentage of Participants Who Experienced a Clinical Exacerbation
Description: Clinical exacerbation is defined as hospitalization because of participant's schizophrenia or requiring change from current antipsychotic or initiation of an adjunctive antipsychotic, 2-point worsening in CGI-S or emergency room visit, deliberate self-injury, emergence of clinically significant suicidal ideation, utilization of treatment team services, violent behavior, requiring an increase in dose of existing antipsychotic as a result of poor symptom control.
Time Frame: Baseline up to Month 24
Population: ITT population included all participants who received medication with at least one post-baseline effectiveness measure. This study was stopped due to futility; care must be exercised in any interpretation of utilization of these data.
Measure: Number; unit: Percentage of participants
Groups:
- Risperidone Long-acting Injection (LAI): Risperidone LAI 25 mg, 37.5 mg or 50 mg intramuscular (injection of a substance into a muscle) injection was administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic was also administered in the first 3 weeks following the dose increase. Duration of treatment was 24 months.
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 86
Percentage of participants | 54.4 | 54.7

3. Secondary Outcome: Time to First Clinical Exacerbation
Description: Time to first clinical exacerbation was calculated over the entire trial duration wherein clinical exacerbation is defined as hospitalization because of participant's schizophrenia or requiring change from current antipsychotic or initiation of an adjunctive antipsychotic, 2-point worsening in CGI-S or emergency room visit, deliberate self-injury, emergence of clinically significant suicidal ideation, utilization of treatment team services, violent behavior, requiring an increase in dose of existing antipsychotic as a result of poor symptom control.
Time Frame: Baseline up to Month 24
Population: ITT population included all participants who received medication with at least one post-baseline effectiveness measure. Here, 'N' signifies number of participants evaluated for this outcome measure. This study was stopped due to futility; care must be exercised in any interpretation of utilization of these data.
Measure: Mean (Standard Error); unit: Months
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 78 | 85
Months | 10.4 (0.80) | 11.2 (0.93)

4. Secondary Outcome: Time in Symptomatic (Having Symptoms) Remission
Description: Time in symptomatic (having symptoms) remission for participants on risperidone was compared with those on oral atypical medication and was calculated over the entire trial duration.
Time Frame: Baseline up to Month 24
Population: Data for this outcome was not computed as it was not defined in terms of the formula for calculation and thus was not included in analysis plan.
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Total Score at Month 24
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210, higher scores indicate worsening.
Time Frame: Baseline and Month 24
Population: ITT population. Here, 'N' signifies number of participants evaluated for this outcome measure. 'n' signifies number of participants who were evaluated for this outcome measure at given timepoint. This study was stopped due to futility; care must be exercised in any interpretation of utilization of these data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 85
Units on a scale
  Baseline (n=79, 85) | 77.6 (17.24) | 76.5 (17.83)
  Change at Month 24: Total score (n=67, 67) | -9.6 (19.80) | -12.4 (21.83)

6. Secondary Outcome: Number of Participants With Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill. Higher scores indicate worsening.
Time Frame: Baseline and End of Study (Month 24 or Early Withdrawal [EW])
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 85
participants
  Baseline: Mild or better (n=79, 85) | 18 | 26
  Baseline: Moderate, marked and severe (n=79, 85) | 61 | 59
  Month 24/EW: Mild or better (n=67, 68) | 36 | 39
  Month 24/EW:Moderate,marked and severe (n=67, 68) | 31 | 29

7. Secondary Outcome: Number of Participants With Clinical Global Impression of Change (CGI-C)
Description: The CGI-C is a assessment of change in global clinical status, defined as a sense of well-being and ability to function in daily activities. CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Higher scores indicate worsening.
Time Frame: End of Study (Month 24 or Early Withdrawal [EW])
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 67 | 68
Participants
  Month 24/EW:At least minimally improved(n= 67,68) | 48 | 38
  Month 24/EW: No change or worse (n=67,68) | 19 | 30

8. Secondary Outcome: Number of Participants With Response to Resource Utilization Questionnaire (RUQ)
Description: This questionnaire included questions asked to participants about any hospitalizations, visits to the emergency room or any other psychiatric treatment received in the previous month. Also the participants and/or primary health care contact or caregiver (or other modality to obtain accurate information) were telephoned on a monthly basis (1 month post Visit 2 through to end of study [Visit 6, Month 24]) by a member of the investigational staff and the resource utilization assessment was conducted over the phone.
Time Frame: Baseline up to Month 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 86
Participants
  Emergency room visits (total reports) | 32 | 29
  Hospital admissions (total reports) | 42 | 32
  Family doctor visits (total reports) | 59 | 58
  Psychologist doctor visit (total reports) | 14 | 13
  Social worker (total reports) | 43 | 44
  Occupational therapist (total reports) | 28 | 30
  Phychiatric day care (total reports) | 19 | 13
  Phychiatrist (total reports) | 74 | 78
  Visit by a home care nurse (total reports) | 15 | 8
  Psychiatric nurse (total reports) | 62 | 58
  Suicide/crisis services (total reports) | 13 | 13
  Outpatient clinic (total reports) | 31 | 36

9. Secondary Outcome: Change From Baseline in Assessment of Quality of Life (AQoL) Score at Month 24
Description: AQoL is defined as an Australian-developed participant delivered quality of life (QoL) instrument consisting of 15-questions in 5 scales measuring illness, independence, social relationships, physical senses and psychological well-being. Each of the 5 scales is calculated based on the answers to 3 questions. Each question is given an answer dependent utility score (0 [worst] to 1 [best] and then these scores are combined using a multiplicative model to get the normalized scale score value, each scale ranging between 0.0 (representing death) and 1.0 (representing full health). The scores for independent living, social relationships, physical senses and psychological well-being are combined to obtain the QoL utility score which refers to the "value" of a health state to the respondent where the lower boundary is -0.04 (representing QoL state worse than death), 0.00 (death equivalent QoL state) and to 1.00 (best possible QoL state)".
Time Frame: Baseline and Month 24
Population: ITT population. Here 'N' signifies number of participants evaluated for this outcome measure and 'n' signifies number of participants who were evaluated for this outcome measure at given timepoint. This study was stopped due to futility; care must be exercised in any interpretation of utilization of these data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 84
Units on a scale
  Baseline: Illness score (n=79,84) | 0.396 (0.2496) | 0.359 (0.2549)
  Change at Month 24: Illness score (n=64,67) | 0.091 (0.3086) | 0.035 (0.3101)
  Baseline: Daily activity score(n=79,83) | 0.811 (0.2312) | 0.872 (0.2156)
  Change at Month 24: Daily activity score(n=64,67) | 0.051 (0.2370) | -0.038 (0.2283)
  Baseline: Social score (n=79,83) | 0.608 (0.2926) | 0.613 (0.3117)
  Change at Month 24: Social score (n=64,66) | 0.060 (0.3143) | 0.025 (0.3474)
  Baseline: Physical score (n=79,83) | 0.872 (0.1437) | 0.916 (0.1022)
  Change at Month 24: Physical score (n=64,67) | 0.065 (0.1581) | 0.020 (0.0919)
  Baseline: Psychological score (n=79,83) | 0.863 (0.1469) | 0.863 (0.1595)
  Change at Month 24: Psychological score (64,67) | 0.015 (0.1677) | 0.023 (0.01527)

10. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) Total Score at Month 24
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
Time Frame: Baseline and End of Study (Month 24 or Early Termination [ET])
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Atypical Antipsychotic
Number analyzed (Participants) | 79 | 84
Units on a scale
  Baseline: (n=79, 84) | 54.2 (13.32) | 55.0 (13.49)
  Change at Month 24/ET: (n=67,68) | 5.2 (17.76) | 8.4 (15.72)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: All participants of the ITT population were included in the safety analysis set. This set thus consisted of 167 participants, 81 randomly assigned to risperidone long-acting injection (LAI), 86 participants randomly assigned to oral antipsychotic treatment.
Arm/Group | Risperidone Long-Acting Injection (LAI) | Oral Atypical Antipsychotic
Serious Adverse Events (participants affected / at risk) | 14/81 | 6/86
Other Adverse Events (participants affected / at risk) | 70/81 | 69/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-Acting Injection (LAI) (N=81) | Oral Atypical Antipsychotic (N=86)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Irritability (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Delusion of grandeur (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Hostility (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-Acting Injection (LAI) (N=81) | Oral Atypical Antipsychotic (N=86)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0
Asthenopia (Eye disorders) | 1 | 0
Blepharopachynsis (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 3 | 4
Crepitations (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 5
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 2
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 0 | 1
Sluggishness (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 2 | 0
External ear cellulitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 2
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Helminthic infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 3 | 4
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 7 | 7
Oral candidiasis (Infections and infestations) | 0 | 1
Oral infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 3 | 2
Tooth infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood alcohol increased (Investigations) | 1 | 1
Blood cholesterol (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 2 | 5
Blood ketone body (Investigations) | 0 | 1
Blood pressure diastolic increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 3
Blood prolactin increased (Investigations) | 3 | 1
Blood triglycerides (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 2 | 3
Blood urea increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 2
Electrocardiogram qt prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 3
Glucose urine present (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 2
Heart rate increased (Investigations) | 0 | 1
High density lipoprotein decreased (Investigations) | 1 | 0
Laboratory test abnormal (Investigations) | 2 | 3
Liver function test abnormal (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 2 | 2
Murphy's sign positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Protein urine (Investigations) | 1 | 0
Semen volume decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 2
Weight increased (Investigations) | 13 | 10
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Central obesity (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 5 | 4
Bradykinesia (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 11 | 10
Dreamy state (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 2 | 0
Dystonia (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 21 | 7
Hypersomnia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 2 | 3
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 3 | 1
Restless legs syndrome (Nervous system disorders) | 4 | 0
Sciatica (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 6
Somnolence (Nervous system disorders) | 5 | 5
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tardive dyskinesia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 5 | 3
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 12 | 11
Anger (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 18 | 14
Apathy (Psychiatric disorders) | 1 | 0
Communication disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delusion (Psychiatric disorders) | 2 | 1
Depressed mood (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 10 | 4
Depressive symptom (Psychiatric disorders) | 2 | 3
Drug abuse (Psychiatric disorders) | 1 | 0
Elevated mood (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 1 | 2
Hallucination, auditory (Psychiatric disorders) | 4 | 1
Hallucination, visual (Psychiatric disorders) | 2 | 0
Ideas of reference (Psychiatric disorders) | 0 | 1
Inappropriate affect (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 21 | 12
Libido decreased (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 3 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0
Orgasm abnormal (Psychiatric disorders) | 0 | 1
Orgasmic sensation decreased (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 1
Persecutory delusion (Psychiatric disorders) | 1 | 0
Pressure of speech (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 4 | 5
Restlessness (Psychiatric disorders) | 3 | 1
Schizophrenia (Psychiatric disorders) | 4 | 3
Sleep disorder (Psychiatric disorders) | 0 | 2
Social avoidant behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Tachyphrenia (Psychiatric disorders) | 1 | 0
Tic (Psychiatric disorders) | 0 | 1
Bladder irritation (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2
Galactorrhoea (Reproductive system and breast disorders) | 2 | 0
Painful erection (Reproductive system and breast disorders) | 1 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 2
Testicular disorder (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 2
Verbal abuse (Social circumstances) | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Removal of foreign body (Surgical and medical procedures) | 0 | 1
Rhinoplasty (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 1
Tooth extraction (Surgical and medical procedures) | 2 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less